CLINICAL TRIAL: NCT03192917
Title: A Prospective Randomized Study Whether Low-energy Extracorporeal Shockwave Therapy (LI-ESWT) Can Increase Erectile Function in Patients After Radical Prostatectomy
Brief Title: Low-energy Extracorporeal Shockwave Treatment for Patients After Radical Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Peter Bill Ladegaard, Student, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S-20170074
Record Dates: First submitted 2017-05-29; First posted 2017-06-20 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Erectile Dysfunction; Post-Op Complication; Prostatic Diseases
Keywords: Shock wave therapy; erectile dysfunction
MeSH Terms: conditions — Erectile Dysfunction; Postoperative Complications; Prostatic Diseases | interventions — salicylhydroxamic acid; Capsules

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active treatment (Experimental): This group of participant will receive low intensity shock wave treatment accounted on their penile shaft once every week for 5 weeks.
  Interventions: Procedure: Low intensity extracorporeal shock wave treatment (LI-ESWT)
- Placebo group (Placebo Comparator): this group of participant will meet up for treatment. The treatment given will be the exact same as the active group, but the transducer used for shock wave treat will me capped, meaning that no shock waves are transmitted to their penis.
  Interventions: Procedure: Low intensity extracorporeal shock wave treatment (LI-ESWT) sham

INTERVENTIONS:
Procedure: Low intensity extracorporeal shock wave treatment (LI-ESWT) — Shock wave treatment with 3000 Hz for 10 min on the penile shaft. This will be done one time a week for five weeks.
  Other Names: Storz Medical AG; DUOLITH® SD1
  Arms: Active treatment
Procedure: Low intensity extracorporeal shock wave treatment (LI-ESWT) sham — A specialized cap can be applied to the chock wave device, which disallow shock waves to transmit through the unit.
  Other Names: DUOLITH® SD1 with cap
  Arms: Placebo group

SUMMARY:
The purpose of this project is to verify the relationship between low intensity shock wave treatment (LI-SWT) and increased scores in self-assessment regarding to erectile function (ED) and sexual intercourse, in patients, who has undergone a radical prostatectomy (RP). The data will be obtained from patients using international accepted sexual questionnaires prior to the LI-SWT and 5, 12 and 24 weeks following treatment.

DETAILED DESCRIPTION:
Extracorporeal shockwave therapy (ESWT) has been used for many years in different fields. In 1980, the clinical use of extracorporeal shockwave lithotripsy as a treatment for stone disease in the upper urinary tract began and proved effective. Throughout the years, ESWT has been modified for use in other specialties, such as in the treatment of gallstones, sialolithiasis and Peyronie's disease. Animal studies have demonstrated neoangiogenesis in myocardial tissue and skin flaps as well as regeneration of nervous tissue. Gotte et al. found that shock waves can, under suitable conditions, lead to non-catalytic synthesis of physiologically relevant quantities of NO. These pioneering findings corroborate our hypothesis that ED due to RP, can likely be treated by LI-SWT.

It is well known that patients radically operated for prostate cancer subsequently develop erectile dysfunction (ED) and /or urinary incontinence. A meta-analysis from 2009 found that the overall erection recovery rate after prostatectomy were 58%, meaning that a certain amount of patients still suffer from ED in the postoperative lifespan.

The investigators want to investigate in a randomized trial whether LI-ESWT is efficient in ED patients, who has undergone RP, regarding to sexual function. These data will be assessed by changes in outcome of sexual questionnaire regarding to sexual function and erection hardness. This hypothesis has previous been tested in a Danish pilot study. The study design was a prospective cohort study with 16 participants all suffering from ED due to nerve sparing RD. The participants received two series of LI-ESWT per week in a 3-week period. The results indicated a gradual increase in erectile function at the 1 month follow up, evaluated by cross matching the IIEF-15 scores before and after treatment. However, the effect was damped off at the last follow up one year later. The pilot study concluded that more research had to be done in a larger population group.

The study design is decided to be a prospective, blinded, randomized placebo-control follow up design. The total enrol of participants are estimated to be sixty-four divided into a placebo group and an active group.

The participants who meet the inclusions criteria (see section below) will be randomly assigned to either a control group (P) or an active group based (V) on a randomization list.

The treatment sessions will take place at the outpatient clinic of the department of urology L, OUH. The shock wave device used for this study is a duolith® SD1 T-Top from Storz Medical (see fig. 2). The device is set at 0.15 mJ/mm2, 5 Hz, with a total of 3000 impulses, and a total energy of 12.8 J per treatment. LI-ESWT will be performed in six positions on the penis (distal, center and proximal part of each cavernous body) and given by a therapist educated for the purpose. The cap used to prevent LI-SWT in the placebo group will be positioned by the Head of the Department to ensure valid blinding.

Prior to the treatment, the participants will be asked to fulfil questionnaires (EHS, IIEF-15 and DAN-PSS) to assess data on lower urinary tract symptoms, sexual dysfunction and erection hardness. At the first treatment session (baseline function), the investigator reviews the questionnaires in cooperation with the participant to ensure no conflicts and misunderstanding in questions.

There will be a total of 5 treatment sessions during a 5-week period. Shortly after treatment, the participants will be asked to fill in the questionnaires once again. The questionnaires will be mailed to the participants home addresses together with a prepaid return envelope and asked to be reposted at 5th, 12th and 24th week respectively.

ELIGIBILITY:
Inclusion Criteria:

* Erectile dysfunction for more than 6 months,
* Time since prostatectomy must be at least 9 month
* At least unilateral nerve-sparing RP.
* Erection Hardness Score (EHS) less than 2 and an Index of Erectile Function (IIEF-5) score less than 17
* Age 20-80 years
* have been in a relationship for more than 3 months.
* Participant can give informed consent.

Exclusion Criteria:

* Men with ED due to other reason than RD (psychogenic, neurological pathology or organic ED etc.)
* Rectal extirpation, radiation therapy to the pelvic area and recovery from any other cancer within the past 5 years are excluded.
* Participants with heart disease prohibiting sexual activity or taking medication with antiandrogens, anticoagulant (apart from aspirin) or systemic use of glucocorticoids within 5 weeks.
* ED treatment within the last 7 days (screening phase), oral medication, vacuum devices, injections.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only men undergone a surgery for prostatectomy will be included in this trial.
Enrollment: 38 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Erection hardness score (EHS) Baseline | 2 weeks prior first treatment
  A five entity questionnaire to review the self-esteem of erection during sexual intercourse. The questionnaire will be mailed to the participants home adresses together with a return envelope.
Erection hardness score first follow up | 5 weeks after last treatment
  A five entity questionnaire to review the self-esteem of erection during sexual intercourse. The questionnaire will be mailed to the participants home adresses together with a return envelope.
Erection hardness score second follow up | 12 weeks after last treatment
  A five entity questionnaire to review the self-esteem of erection during sexual intercourse. The questionnaire will be mailed to the participants home adresses together with a return envelope.
Erection hardness score third follow up | 24 weeks after last treatment.
  A five entity questionnaire to review the self-esteem of erection during sexual intercourse. The questionnaire will be mailed to the participants home adresses together with a return envelope.

SECONDARY OUTCOMES:
The International index of erection function (IIEF-5) baseline | 2 weeks prior first treatment
  A fifteen item questionnaires to access data on erection function. Only question 1-5 will be used in for data interpretation. These item is also called til erection function domain (EF domain)
The International index of erection function (IIEF-5) first follow up | 5 weeks after last treatment
  A fifteen item questionnaires to access data on erection function. Only question 1-5 will be used in for data interpretation. These item is also called til erection function domain (EF domain)
The International index of erection function (IIEF-5) second follow up | 12 weeks after last treatment
  A fifteen item questionnaires to access data on erection function. Only question 1-5 will be used in for data interpretation. These item is also called til erection function domain (EF domain)
The International index of erection function (IIEF-5) third follow up | 24 weeks after last treatment
  A fifteen item questionnaires to access data on erection function. Only question 1-5 will be used in for data interpretation. These item is also called til erection function domain (EF domain)

OTHER OUTCOMES:
Danish Prostate Symptoms Scoring scheme (DAN-PSS) | 2 weeks prior first treatment
  A 12 item questionsaires regarding lower urinary tracts symptoms. Used to access whether there is any additional effects of the treatment
Danish Prostate Symptoms Scoring scheme (DAN-PSS) | 24 weeks after last treatment
  A 12 item questionsaires regarding lower urinary tracts symptoms. Used to access whether there is any additional effects of the treatment
Pain sensation | first treatment
  All participants are asked by the investigator, shortly after treatment, if there were any pain sensations during the application of shockwaves. This will be notified on a scheme.
Pain sensation | second treatment (1 week after first treatment)
  All participants are asked by the investigator, shortly after treatment, if there were any pain sensations during the application of shockwaves. This will be notified on a scheme.
Pain sensation | third treatment (2 week after first treatment)
  All participants are asked by the investigator, shortly after treatment, if there were any pain sensations during the application of shockwaves. This will be notified on a scheme.
Pain sensation | fourth treatment (3 week after first treatment)
  All participants are asked by the investigator, shortly after treatment, if there were any pain sensations during the application of shockwaves. This will be notified on a scheme.
Pain sensation | fifth treatment (4 week after first treatment)
  All participants are asked by the investigator, shortly after treatment, if there were any pain sensations during the application of shockwaves. This will be notified on a scheme.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Lund, MD professor, Study Chair — Department of Urology
Locations (1):
- Odense University Hospital (OUH), Odense, Fyn, Denmark

IPD SHARING:
Plan to Share IPD: No